CLINICAL TRIAL: NCT02495870
Title: The Acute Effects of Low Temperature for Long Time Heat Treatment of Pork Semitendinosus on Satiety
Acronym: SAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Meat Research Institute (Other)
Responsible Party: Principal Investigator, Anne Birgitte Raben, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SAPO 2A
Record Dates: First submitted 2014-11-10; First posted 2015-07-13 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Pork Meat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pork, 58°C, 72 minutes (Experimental): Pork muscle (semitendinosus) sous-vide cooked at 58°C for 72 minutes
  Interventions: Other: Pork
- Pork, 58°C, 17 hours (Experimental): Pork muscle (semitendinosus) sous-vide cooked at 58°C for 17 hours
  Interventions: Other: Pork
- Meat balls, 58°C, 17 hours (Experimental): Meat balls made from pork Semitendinosus. Sous-vide cooked at 58°C for 17 hours
  Interventions: Other: Pork
- Pork, 160°C (until 58°C in core) (Active Comparator): Pork muscle (semitendinosus) oven cooked at 160°C until 58° in core.
  Interventions: Other: Pork

INTERVENTIONS:
Other: Pork

SUMMARY:
Cooking meat at low temperatures for prolonged times is widely used among chefs and in food service due to the possibility to obtain a consistent and appealing eating quality. The method is generally termed low-temperature long-time (LTLT) cooking. In LTLT cooking, meat is vacuum-packed and heated at temperatures between 50°C and 65°C in a water bath for several hours. LTLT has several benefits - improved tenderness and juiciness, less cooking loss, better vitamin retention and uncompromised food safety.

A recent PhD thesis concluded that one of the mechanisms behind the changes in eating quality during LTLT cooking was due to the proteolytic degradation in the muscle tissue. The activity of proteolytic enzymes has shown to be dependent on heating temperature and time where the cathepsins were found to remain active during heat treatment. At 58°C the cathepsin B+L activity is increased compared to 48°C and 53°C and at 55°C compared to 25°C, 40°C and 70°C. A prolonged heating time of 17 hours at 58°C has also shown to increase cathepsin B+L activity. The proteolytic degradation results in the occurrence of peptides and amino acids such as tryptophan, tyrosine, leucine and histidine which could lead to a faster degree of satiety when consumed.

According to the aminostatic hypothesis by Mellinkoff, a rise in plasma amino acids elicited by protein ingestion could assist in the suppression of food intake and the onset of satiety.

The investigators therefore hypothesize that the ingestion of LTLT cooked pork would induce a faster satiety response due to the higher availability of peptides and amino acids prior to digestion. An acute meal study will elucidate this. LTLT cooking will be performed by the "cook-chill" method to mimic real life where meat is rapidly chilled after heat treatment, stored at 0-2°C and reheated and browned prior to serving.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Healthy men
* Ages between 18 and 60 years
* BMI between 18.5 and 30 kg/m2
* Pork eaters

Exclusion Criteria:

* Any food allergy, dislike or special diet of relevance to the study (e.g. vegetarian)
* Daily use of prescription medicine or over-the-counter drugs affecting appetite, energy expenditure or protein metabolism
* Use of dietary supplements (including protein supplement, powders, shakes) up to 1 month before the first meal test
* Irregular eating schedule (e.g. skipping breakfast)
* Self-reporting currently dieting or having lost/gained significant amount of weight (±3 kg) in the previous 3 months
* Any known chronic diseases (e.g. cancer, heart disease, diabetes, neurological disorders)
* Vigorous physical activity more than 10 hours/week
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes) (>10 cigarettes per day)
* Participants who work in appetite or feeding related areas
* Participation in other intervention studies
* Participants not able to comply with the study protocol as judged by study personnel

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake | 180 min
  the primary outcome is measured 180 min after test meal is consumed

SECONDARY OUTCOMES:
VAS scores for appetite (hunger, satiety, fullness, prospective consumption) | every 30 min at time points 15, 45, 75, 105, 135, 165, 195 min from termination of the test meal.
  The secondary endpoints are measured every 30 minute after the test meal is consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Meat Research Institute, Taastrup, Denmark